CLINICAL TRIAL: NCT07389538
Title: Promoting Safe Medication Practices in the Classroom: Medicación Con-Ciencia
Brief Title: Promoting Safe Medication Practices in the Classroom
Acronym: MedConCiencia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Ministerio de Ciencia, Innovación y Universidades (Unknown)
Responsible Party: Principal Investigator, María Correa-Rodríguez, Associate Professor, Universidad de Granada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4384/CEIH/2024
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Self Medication
Keywords: Health Literacy; Adolescent; Quality of Life; Self Medication; Artificial Intelligence; Education
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Longitudinal quasi-experimental clinical trial with a non-randomized control group in young people aged 15 to 24 years, designed to assess self-medication practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group consisted of participants who were absent during the intervention but completed the post-intervention questionnaire.
- Educational intervention (Experimental): Group receiving the structured educational program focused on the appropriate use of medications and the prevention of errors associated with self-medication.
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — The intervention will consist of a structured educational program focused on the appropriate use of medications and the prevention of errors associated with self-medication.
  Arms: Educational intervention

SUMMARY:
Self-medication has traditionally been defined as the consumption of medicines, herbs, and home remedies on one's own initiative or on the advice of another person, without consulting a doctor. In Spain, the consumption of non-prescription drugs is quite widespread among young people, since more than half of them have used medications without a medical prescription in the last year.

This high prevalence of self-medication among Spanish youth seems to be driven by various factors that encourage this practice. These include the increase in over-the-counter medications, delays in obtaining appointments at health centers, the influence of common family self-care practices, and the population's greater knowledge of and interest in health-related issues.

Inappropriate use of medications constitutes a public health problem and can cause significant risks to users' health, such as adverse reactions, drug resistance, and complications in diagnosing diseases, since it can lead to the masking of symptoms, as well as an increase in morbidity.

However, not all self-medication practices are harmful. Responsible self-medication refers to the use of over-the-counter medications (without a prescription) to treat common and mild symptoms (e.g., fever, mild pain, colds) for a reasonable period of time (two to three days, after which a doctor should be consulted if no improvement occurs). The benefits of responsible self-medication include convenience for the patient, reinforcement of personal autonomy through self-care, reduction of healthcare professionals' workload, and decreased costs to the healthcare system. In this regard, responsible self-medication not only provides individual and collective benefits but also promotes the development of personal autonomy, a key factor influencing young people's tendency to self-medicate. Attitudes toward autonomous medication use in young people are influenced by individual variables such as emotional regulation, family habits, peer influence, quality of life, and the use of other substances.

Given that these factors-greater access to medications, delays in healthcare access, family self-care practices, and individual psychosocial characteristics-appear to drive self-medication behaviors among youth, it is hypothesized that an educational intervention developed with the support of artificial intelligence, and focused on the responsible and safe use of medications, will improve young people's knowledge and attitudes toward self-medication. By targeting both knowledge and attitudes, the intervention aims to strengthen responsible practices while fostering autonomy and informed decision-making in medication use.

DETAILED DESCRIPTION:
The present study is grounded in the premise that widespread lack of knowledge regarding the appropriate use of medications represents a relevant educational and public health problem that should be addressed from early stages of life. Accordingly, the primary objective of this study is to improve health literacy related to responsible self-medication among young people.

To achieve this objective, a longitudinal quasi-experimental clinical trial with a non-randomized control group was designed. The study will include young individuals aged 15 to 24 years recruited from secondary schools, vocational training programs, and undergraduate degree programs in the province of Granada. Data will be collected at two predefined time points: a baseline assessment conducted prior to the intervention (pre-intervention) and a follow-up assessment performed 6 to 9 months after the intervention (post-intervention).

At both assessment points, participants will independently complete a structured questionnaire collecting information on sociodemographic characteristics, self-medication practices, knowledge and attitudes toward self-medication, as well as physical and psychosocial factors. The outcome measures will be primarily assessed using validated instruments, including the Kidscreen-27 (Screening for Health-Related Quality of Life in Children and Adolescents, 27-item version) and the QAR-LS questionnaires (Risk Self-Medication Questionnaire focused on Health Literacy), ensuring the reliability and validity of the data collected.

Participants will be allocated to one of two study groups: an intervention group and a control group with a smaller sample size. Due to the non-randomized nature of the study, allocation to the control group will be determined by participants' absence during the implementation of the educational intervention. Participants in the control group will not receive the intervention but will complete the post-intervention assessment, allowing for between-group comparisons.

The intervention will consist of a structured educational program focused on the appropriate use of medications and the prevention of errors associated with self-medication. The program will be delivered face-to-face in participating educational institutions during regular school hours and within classroom settings, with an estimated duration of approximately two hours. The intervention will integrate theoretical and practical components organized into four workshops.

To enhance intervention fidelity and ensure suitability for the target population, artificial intelligence-based tools will be employed to adapt educational materials to participants' age and to language accessible to the general population. In addition, graphic and audiovisual resources, together with gamification strategies, will be incorporated to promote engagement and facilitate learning. As a complementary component, a gamified virtual escape room will be developed to encourage safe medication-use practices and to prevent risk behaviors among young people, thereby extending the potential reach of the intervention to young populations nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include being a student at secondary education institutions, vocational training programs, or undergraduate degree programs in the province of Granada, and being between 15 and 24 years of age.

Exclusion Criteria:

* Exclusion criteria will include: lack of informed consent from the participant or their legal guardians in the case of minors, and the presence of barriers that prevent proper understanding of the questionnaires and activities to be carried out (e.g., language barriers, intellectual disability, etc.).

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Risk Self-Medication Questionnaire focused on Health Literacy (QAR-LS) | Data will be collected at baseline and again 6-9 months after the intervention.
  The Risk Self-Medication Questionnaire focused on Health Literacy (QAR-LS) provides scores ranging from 35 to 175 points, where higher scores indicate a greater risk related to inadequate or unsafe self-medication practices.

SECONDARY OUTCOMES:
Health-related quality of life (Kidscreen-27) | Data will be collected at baseline and again 6-9 months after the intervention.
  The KIDSCREEN-27 (Screening for Health-Related Quality of Life in Children and Adolescents, 27-item version) consists of 27 items covering five dimensions: physical well-being, psychological well-being, autonomy and parent relations, social support and peers, and school environment. When summed, total raw scores may range from 27 to 135, although interpretation is typically based on dimension scores or standardized T-scores. Higher scores reflect better health-related quality of life.
Problem-focused coping styles (COPE-28) | Data will be collected at baseline and again 6-9 months after the intervention.
  The COPE-28 (Coping Orientation to Problems Experienced, 28-item version) consists of 28 items rated on a 4-point Likert scale. When summed, total scores range from 28 to 112, although interpretation is typically based on its subscales. Higher scores indicate greater use of the coping strategies assessed.
  The instrument includes 14 two-item subscales measuring specific coping responses, such as active coping, planning, seeking emotional or instrumental support, positive reframing, acceptance, humor, religion, self-distraction, denial, venting, substance use, behavioral disengagement, and self-blame. These can be grouped into broader domains (e.g., problem-focused, emotion-focused, dysfunctional coping).

CONTACTS AND LOCATIONS:
Overall Officials: María Correa-Rodríguez, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramírez Puerta, D., Larrubia Muñoz, O., Escortell Mayor, E., & Martínez Martínez, R. (2006). La automedicación responsable, la publicidad farmacéutica y su marco en la Atención Primaria. SEMERGEN, Soc. Esp. Med. Rural Gen. (Ed. impr.), 117-124.
- [Background] Morán, C., Landero, R., & González, M. T. (2010). COPE-28: un análisis psicométrico de la versión en español del Brief COPE. Universitas Psychologica, 9(2), 543-552.
- [Background] Kidscreen Group (2004). Estudio europeo de salud y bienestar de niños/as y adolescentes. Cuestionario para chicos y chicas de 8 a 18 años. https://www.kidscreen.org/english/questionnaires/kidscreen-27/
- [Background] Barreto, M. A. F., Negreiros, F. D. D. S., Cestari, V. R. F., Sampaio, H. A. C., & Moreira, T. M. M. (2024). Evidence of validity of the Risk Self-Medication Questionnaire focused on Health Literacy. Revista brasileira de enfermagem, 77(3), e20230386. https://doi.org/10.1590/0034-7167-2023-0386
- [Background] Baracaldo-Santamaría, D., Trujillo-Moreno, M. J., Pérez-Acosta, A. M., Feliciano-Alfonso, J. E., Calderon-Ospina, C. A., & Soler, F. (2022). Definition of self-medication: a scoping review. Therapeutic advances in drug safety, 13, 20420986221127501. https://doi.org/10.1177/20420986221127501